CLINICAL TRIAL: NCT02013817
Title: CHAIROS - Effect of Early Brief Intensification by Chemoimmunotherapy With FCR Followed by FR and Rituximab Maintenance on Clinical Response in Chemo-naïve Patients With B-CLL
Brief Title: CHAIROS Study A Study of MabThera/Rituxan (Rituximab) Maintenance Therapy in Patients With B-Cell Chronic Lymphocytic Leukemia (CLL) Naive to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18434
Record Dates: First submitted 2013-12-03; First posted 2013-12-17 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; fludarabine; Cyclophosphamide

ARMS (1):
- MabThera/Rituxan (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: fludarabine; Drug: cyclophosphamide

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — Every 4 weeks for 6 cycles of induction, followed by maintenance therapy every 3 months x 8
Drug: fludarabine — Every 4 weeks, 6 cycles
Drug: cyclophosphamide — Every 4 weeks, 3 cycles

SUMMARY:
This study will evaluate the efficacy and safety of intense combination treatment including MabThera/Rituxan (rituximab), followed by MabThera/Rituxan maintenance therapy in patients with B-cell CLL who are naive to chemotherapy. The anticipated time on study treatment is 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* B-cell CLL
* No previous chemotherapy, radiotherapy, or immunotherapy

Exclusion Criteria:

* Reduced organ function, or bone marrow dysfunction not due to CLL
* Patients with a history of other malignancies within 2 years prior to study entry, except for adequately treated cancer in situ of the cervix, or basal or squamous cell skin cancer
* Patients with a history of severe cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-10-11 (Actual); Primary Completion 2012-09-24 (Actual); Study Completion 2012-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (8):
- Austria (8):
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Innere Medizin Abt. Für Hämatologie & Onkologie, Innsbruck
  - LKH Hochsteiermark; Abt. für Innere Medizin, Leoben
  - Kh Der Barmherzigen Schwestern; Interne I X, Linz
  - A.Ö. Krankenhaus Der Elisabethinen Linz; I. Interne Abt., Linz
  - Kepler Universitätskliniken GmbH - Med Campus III; I. Medizinische Abteilung, Linz
  - Landeskrankenhaus Rankweil; Interne E, Rankweil
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Klinikum Kreuzschwestern Wels; Iii. Interne Abt., Wels

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab, Fludarabine, Cyclophosphamide: Induction Phase Cycle 1 (4-week cycle): Participants received fludarabine 25 milligrams per square meter (mg/m^2) intravenously (IV) and cyclophosphamide 250 mg/m^2 IV on Days 1-3 and rituximab 375 mg/m^2 IV on Day 4. Induction Phase Cycles 2 and 3 (4-week cycles): Participants received rituximab 500 mg/m^2 IV on Day 1 and fludarabine 25 mg/m^2 IV and cyclophosphamide 250 mg/m^2 IV on Days 1-3 Induction Phase Cycles 4 to 6 (4-week cycles): Participants received rituximab 500 mg/m^2 IV on Day 1 and fludarabine 25 mg/m^2 IV on Days 1-5. Maintenance Phase (Cycles 1-8; 12-week cycles): 8 weeks after the end of the last induction cycle, participants received maintenance therapy with rituximab 375 mg/m^2, IV once every 12 weeks for a total of 8 infusions (maximum 2 years).
Period: Overall Study
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Started | 43
Completed | 16
Not Completed | 27
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 4
Not completed — Death | 2
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) population: all participants who received at least one dose of study medication.
Groups:
- Rituximab, Fludarabine, Cyclophosphamide: Induction Phase Cycle 1 (4-week cycle): Participants received fludarabine 25 mg/m^2 IV and cyclophosphamide 250 mg/m^2 IV on Days 1-3 and rituximab 375 mg/m^2 IV on Day 4. Induction Phase Cycles 2 and 3 (4-week cycles): Participants received rituximab 500 mg/m^2 IV on Day 1 and fludarabine 25 mg/m^2 IV and cyclophosphamide 250 mg/m^2 IV on Days 1-3 Induction Phase Cycles 4 to 6 (4-week cycles): Participants received rituximab 500 mg/m^2 IV on Day 1 and fludarabine 25 mg/m^2 IV on Days 1-5. Maintenance Phase (Cycles 1-8; 12-week cycles): 8 weeks after the end of the last induction cycle, participants received maintenance therapy with rituximab 375 mg/m^2, IV once every 12 weeks for a total of 8 infusions (maximum 2 years).
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Clinical Response of Clinical Remission (CR)
Description: Best clinical response was determined according to the National Cancer Institute (NCI) Clinical and Clinical plus (+) Radiological evaluations by central response assessment. Assessment of response was performed according to the NCI revised guidelines for the diagnosis and treatment of chronic lymphocytic lymphoma (CLL) with additional computerized tomography (CT) scan evaluation of lymphadenopathy. Per NCI guidelines, CR requires all of the following criteria at least 2 months after the last treatment: no lymphadenopathy (Ly)/ hepatomegaly/ splenomegaly/constitutional symptoms; neutrophils greater than (>)1500 per microliter (/µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11.0 grams per deciliter (g/dL), lymphocytes (LC) (less than) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC.
Time Frame: Weeks 1, 5, 9, 12, 13, 17, 21 and 24
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Number analyzed (Participants) | 38
percentage of participants
  NCI Clinical | 73.7 [56.9 to 86.6]
  NCI Clinical (including CRu, CRi) | 94.7 [82.3 to 99.4]
  NCI Clinical + Radiological | 63.2 [46.0 to 78.2]
  NCI Clinical + Radiological (including CRu, CRi) | 78.9 [62.7 to 90.4]

2. Secondary Outcome: Percentage of Participants With the Best Clinical Response by Visit (Clinical Assessment)
Description: Best clinical response was determined according to the NCI clinical evaluation and through radiological assessment. CR, CRi, CRu, partial remission (PR), partial remission with toxicity associated (PRTox), progressive disease (PD), and stable disease (SD) were evaluated. Assessment of response was performed according to the NCI revised guidelines for the diagnosis and treatment of CLL with additional CT scan evaluation of lymphadenopathy during the treatment period (Radiological). Response assessment for interim (Week 12), end of induction (Week 24) and at Final Staging (4 weeks after last maintenance dose). Last observation carried forward (LOCF) method was used for missing data. Percentages are based on the number of nonmissing observations within each stratum.
Time Frame: Weeks 12 and 24 and at Final Staging (Week 4 after last maintenance dose)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Number analyzed (Participants) | 43
percentage of participants
  CR, Week 12 | 41.9 [27.0 to 57.9]
  CRu, Week 12 | 16.3 [6.8 to 30.7]
  CRi, Week 12 | 16.3 [6.8 to 30.7]
  PR, Week 12 | 11.6 [3.9 to 25.1]
  PRTox, Week 12 | 2.3 [0.1 to 12.3]
  SD, Week 12 | 0.0 [0.0 to 8.2]
  PD, Week 12 | 0.0 [0.0 to 8.2]
  Not evaluable, Week 12 | 11.6 [3.9 to 25.1]
  CR, Week 24 | 30.2 [17.2 to 46.1]
  CRu, Week 24 | 11.6 [3.9 to 25.1]
  CRi, Week 24 | 37.2 [23.0 to 53.3]
  PR, Week 24 | 9.3 [2.6 to 22.1]
  PRTox, Week 24 | 0.0 [0.0 to 8.2]
  SD, Week 24 | 0.0 [0.0 to 8.2]
  PD, Week 24 | 0.0 [0.0 to 8.2]
  Not evaluable, Week 24 | 11.6 [3.9 to 25.1]
  CR, Final staging | 60.5 [44.4 to 75.0]
  CRu, Final staging | 7.0 [1.5 to 19.1]
  CRi, Final staging | 11.6 [3.9 to 25.1]
  PR, Final staging | 7.0 [1.5 to 19.1]
  PRTox, Final staging | 0.0 [0.0 to 8.2]
  SD, Final staging | 0.0 [0.0 to 8.2]
  PD, Final staging | 2.3 [0.1 to 12.3]
  Not evaluable, Final staging | 11.6 [3.9 to 25.1]

3. Secondary Outcome: Percentage of Participants With the Best Clinical Response by Visit (Clinical + Radiological Assessment)
Description: Best clinical response was determined according to the NCI clinical evaluation and through radiological assessment. CR, CRi, CRu, PR, PRTox, PD, and SD were evaluated. Assessment of response was performed according to the NCI revised guidelines for the diagnosis and treatment of CLL with additional CT scan evaluation of lymphadenopathy during the treatment period (Radiological). Response assessment for interim (Week 12), end of induction (Week 24) and at Final Staging (4 weeks after last maintenance dose). LOCF method was used for missing data. Percentages are based on the number of nonmissing observations within each stratum.
Time Frame: Weeks 12 and 24 and at Final Staging (Week 4 after last maintenance dose)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Number analyzed (Participants) | 43
percentage of participants
  CR, Week 12 | 30.2 [17.2 to 46.1]
  CRu, Week 12 | 4.7 [0.6 to 15.8]
  CRi, Week 12 | 7.0 [1.5 to 19.1]
  PR, Week 12 | 30.2 [17.2 to 46.1]
  PRTox, Week 12 | 9.3 [2.6 to 22.1]
  SD, Week 124 | 7.0 [1.5 to 19.1]
  PD, Week 12 | 0.0 [0.0 to 8.2]
  Not evaluable, Week 12 | 11.6 [3.9 to 25.1]
  CR, Week 24 | 23.3 [11.8 to 38.6]
  CRu, Week 24 | 7.0 [1.5 to 19.1]
  CRi, Week 24 | 30.2 [17.2 to 46.1]
  PR, Week 24 | 14.0 [5.3 to 27.9]
  PRTox, Week 24 | 7.0 [1.5 to 19.1]
  SD, Week 24 | 7.0 [1.5 to 19.1]
  PD, Week 24 | 0.0 [0.0 to 8.2]
  Not evaluable, Week 24 | 11.6 [3.9 to 25.1]
  CR, Final staging | 48.8 [33.3 to 64.5]
  CRu, Final staging | 7.0 [1.5 to 19.1]
  CRi, Final staging | 7.0 [1.5 to 19.1]
  PR, Final staging | 11.6 [3.9 to 25.1]
  PRTox, Final staging | 2.3 [0.1 to 12.3]
  SD, Final staging | 2.3 [0.1 to 12.3]
  PD, Final staging | 9.3 [2.6 to 22.1]
  Not evaluable, Final staging | 11.6 [3.9 to 25.1]

4. Secondary Outcome: Time to Next Treatment - Percentage of Participants With an Event
Description: Time to next treatment was calculated as the number of days from either discontinuation of the study drug or the administration of the last dose, until the participants needed next treatment.
Time Frame: Weeks 1, 5, 9, 12, 13, 17, 21 and 24 and every 8 weeks for 64 Weeks and every 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Number analyzed (Participants) | 43
percentage of participants | 37.2

5. Secondary Outcome: Time to Next Treatment - Time to Event
Description: as for outcome 4
Time Frame: Weeks 1, 5, 9, 12, 13, 17, 21 and 24 and every 8 weeks for 64 Weeks and every 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Number analyzed (Participants) | 43
days | 423.3 (398.5)

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: AEs were recorded from the date of first medication administration until 28 days after the last trial medication.
Time Frame: Day 1 of Cycles 1, 2, 3, 4, 5, and 6 to 28 days after the last trial medication.
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Number analyzed (Participants) | 43
percentage of participants
  Any AE | 100
  Related AE | 93.0
  Severe AE | 76.7
  SAE | 62.8
  Pregnancy | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the date of first medication administration until 28 days after the last trial medication.
Description: Number and percentage of subjects with at least one AE/SAE starting during study until within 28 days after the last trial medication by stem organ class and preferred term.
Arm/Group | Rituximab, Fludarabine, Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 30/43
Other Adverse Events (participants affected / at risk) | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab, Fludarabine, Cyclophosphamide (N=43)
Bronchitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia primary atypical (Infections and infestations) | 1
Postoperative infection (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Urninary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Pyrexia (General disorders) | 5
Chest pain (General disorders) | 2
Drug intolerance (General disorders) | 1
General physical health deterioration (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Capillary leak syndrome (Vascular disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cataract operation (Surgical and medical procedures) | 1
Prostatic operation (Surgical and medical procedures) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Ateriogram coronary (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Encephalitis herpes (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab, Fludarabine, Cyclophosphamide (N=43)
Leukopenia (Blood and lymphatic system disorders) | 20
Neutropenia (Blood and lymphatic system disorders) | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Anaemia (Blood and lymphatic system disorders) | 13
Lymphopenia (Blood and lymphatic system disorders) | 14
Haemolysis (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Nasopharyngitis (Infections and infestations) | 8
Rhinitis (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 4
Herpes simplex (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Fungal infection (Infections and infestations) | 2
Infection (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 3
Bronchitis bacterial (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 2
Fungal rash (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Omphalitis (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Postoperative infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 1
Pyrexia (General disorders) | 7
Fatigue (General disorders) | 8
Oedema peripheral (General disorders) | 4
Chest pain (General disorders) | 1
Chills (General disorders) | 3
Influenza like illness (General disorders) | 3
Pain (General disorders) | 3
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Bowel movement irregularity (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia exertional (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Oedema genital (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Visual acuity reduced (Eye disorders) | 2
Burnout syndrome (Psychiatric disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 7
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Carotid artery stenosis (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Convulsions local (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Sensory loss (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 3
Circulatory collapse (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Vein pain (Vascular disorders) | 1
Venous insufficiency (Vascular disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 2
Lactose intolerance (Metabolism and nutrition disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Food allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Neck injury (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dysuria (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Micturition disorder (Renal and urinary disorders) | 1
Depression (Psychiatric disorders) | 1
Bronchitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.